CLINICAL TRIAL: NCT00427076
Title: Treatment With Cotrimoxazole vs. Vancomycin for Infections Caused by Methicillin-resistant Staphylococcus Aureus: Randomized Controlled Trial
Brief Title: Cotrimoxazole Versus Vancomycin for Invasive Methicillin-resistant Staphylococcus Aureus Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mical Paul, Dr., Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol V.3, dated 01.06.09
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Staphylococcal Infections; Meningitis; Sepsis; Pneumonia
Keywords: vancomycin; cotrimoxazole; trimethoprim/ sulfamethoxazole; methicillin-resistant Staphylococcus aureus; Health care association infections; MRSA bacteremia or other microbiologically documented MRSA infections (defined clinically by CDC criteria); Suspected neurosurgical meningitis; Sepsis during hemodialysis, catheter-associated and catheter-related infections; Ventilator-associated pneumonia; Surgical site infection in the presence of a foreign body
MeSH Terms: conditions — Staphylococcal Infections; Meningitis; Sepsis; Pneumonia; Catheter-Related Infections; Pneumonia, Ventilator-Associated | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Cotrimoxazole
  Interventions: Drug: Cotrimoxazole
- B (Active Comparator): Vancomycin
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Cotrimoxazole — Cotrimoxazole arm: intravenous cotrimoxazole 4 amp (320 mg trimethoprim/ 1600 mg sulfamethoxazole) diluted in 500 ml D5W or N.S. Q 12 hours. Patients intolerant of volume overload will be given the same dose in 250ml D5W (as in the current recommendations used in the hospital). The dose was selected basing on the existing randomized controlled trial and a pharmacokinetic study . 21 For patients with GFR< 30 the dosage interval will be increased to 4 amp (320 mg trimethoprim/ 1600 mg sulfamethoxazole) diluted in 500 ml D5W or N.S. Q 24 hours. 22 Patients on peritoneal dialysis will be given 2 amp (160 mg trimethoprim/ 800 mg sulfamethoxazole) Q 48 hours. Patients with acute renal failure treated with hemodialysis will be given the 2 amp (160 mg trimethoprim/ 800 mg sulfamethoxazole) after dialysis. Patients on continuous hemofiltration for acute renal failure will be administered the dose for GFR<30.
  Arms: A
Drug: Vancomycin — intravenous vancomycin 1gr Q 12 hours. Adjustment to creatinine clearance: GFR 10-50 1 gr Q 24-96 hours, GFR <10 1gr Q 4-7 days.
  Arms: B

SUMMARY:
Methicillin-resistant Staphylococcus aureus (SA) is a major pathogen causing mainly health-care associated infections and, lately, also community acquired infections. Few treatment choices exist to treat these infections. The currently recommended antibiotics for these infections are glycopeptides (vancomycin or teicoplanin). Glycopeptide treatment hs several disadvantages. It is a last resort antibiotic family that should be reserved for the future; Vancomycin is less effective that beta-lactam drugs for SA infections susceptible to both agents; treatment can only be given intravenously; and use of vancomycin has led to the development of SA strains with partial or complete resistance to vancomycin. Cotrimoxazole is an old antibiotic active against most strains of MRSA, depending on local epidemiology.

Study hypothesis: The purpose of this study is to show that cotrimoxazole is as effective as treatment with vancomycin for invasive MRSA infections.

We plan a randomized controlled trial comparing treatment with cotrimoxazole vs. vancomycin for invasive MRSA infections. The primary efficacy outcome we will assess will be Improvement or cure with or without antibiotic modifications, defined as: survival at 7 days post randomization with resolution of fever (<38 for two consecutive days) and resolution of hypotension (>90 systolic without need for vasopressor support); and physician's assessment that the primary infection was improved or cured. The primary safety outcome will be all-cause 30-day survival.

DETAILED DESCRIPTION:
Staphylococcus aureus (SA) is a major pathogen causing community-acquired and health-care associated infections. In hospitals, SA infections are associated with a significant burden; in-hospital mortality during the last 15 years following SA bacteremia in Beilinson hospital was 38% and did not decrease in recent years. Resistance to beta-lactams is widely prevalent in hospitals (57% of all SA isolates causing bacteremia at our center). The drug of choice currently recommended for these infections is a glycopeptide (vancomycin or teicoplanin).

Cotrimoxazole (trimethoprim-sulfamethoxazole) is a relatively 'old' drug commonly used for urinary tract infections. Invitro, it is active against SA, including methicillin-resistance Staphylococcus aureus (MRSA) strains and its activity against SA is bactericidal. Trimethoprim alone is bactericidal against SA, while sulphamethoxazole alone is relatively inactive and their combination is synergistic both in-vitro and invivo. The prevalence of cotrimoxazole-susceptible SA varies locally. At our center, 97% of SA strains causing bacteremia in 2004 were susceptible to cotrimoxazole. Community-acquired MRSA, prevalent in the United States as a cause for severe skin and soft tissue infections, has not been described in Israel.

Several reasons exist to search for antibiotics other than vancomycin for MRSA infections. Vancomycin is less effective that beta-lactam drugs for SA infections susceptible to both agents. It is the last resort antibiotic for MRSA infections out of the currently recommended bactericidal antibiotics for invasive infections. Use of vancomycin has led to the development of SA strains with partial or complete resistance to vancomycin (VISA and VRSA, respectively). Vancomycin use is associated with the appearance of vancomycin-resistant enterococcus (VRE) species. Nosocomial infections with VISA and VRE are difficult to treat and may spread rapidly in the hospital. 10 Finally, vancomycin cannot be administered orally.

Limited evidence supports the efficacy of cotrimoxazole for MRSA infections, with paucity of data for high-burden invasive infections. Cotrimoxazole is probably inferior to vancomycin for methicillin-susceptible SA. ; thus we may infer indirectly its inferiority to methicillin and drugs alike for MRSA infections. Cotrimoxazole may be less effective than glycopeptides and oxacillin for left-sided endocarditis. No evidence exists to support the use of cotrimoxazole empirically for the treatment of suspected SA infections in the hospital.

We plan an open label single-center pragmatic randomized controlled trial to compare cotrimoxazole to vancomycin. We will include patients with documented or highly suspected MRSA infections, according to pre-defined risk factors. We chose to target this patient population to assess the efficacy of cotrimoxazole both empirically and for documented infections.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* providing signed informed consent or, if unable, having a legal guardian or a caretaker that will sign informed consent
* Patients with documented MRSA infections:
* MRSA bacteremia
* Other microbiologically documented MRSA infections defined as a clinical source of infection (CDC criteria) plus microbiological documentation of MRSA from the source of infection
* Patients with highly probable MRSA infections, prior to microbiological documentation of the pathogen:
* Suspected neurosurgical meningitis (including VP-shunt meningitis)
* Sepsis during hemodialysis
* Ventilator-associated pneumonia with prior antibiotic treatment within 48 hours
* Catheter-related or suspected catheter-related infections
* Surgical site infection in the presence of a foreign body

Exclusion Criteria:

Exclusion before randomization:

* Previous antibiotic treatment directed against MRSA >48 hours (including vancomycin, fucidic acid, rifampicin or cotrimoxazole)
* Known allergy to either study drug
* Acute leukemia and/ or BMT with neutropenia <500/mm3 or <1000/mm3 and expected to decrease below 500/mm3
* Pregnancy, lactation
* Previous enrollment in this study
* Concurrent participation in another trial

Exclusions after randomization:

* Documented Staphylococcal infection resistant to cotrimoxazole or VISA or VRSA
* Documented MSSA
* Documented left-sided endocarditis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2007-06; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Primary efficacy: Improved or cure with or without antibiotic modifications, defined as: survival at 7 days post randomization with resolution of fever and resolution of hypotension | 7 days
Primary safety: 30-day all cause mortality | 30 days

SECONDARY OUTCOMES:
Improved or cure without antibiotic modifications | 7 days
Modification of the anti-staphylococcal treatment within 1 week of treatment onset for perceived failure of therapy | 7 days
Survival at 7 days post randomization without the need for modification of the anti-staphylococcal antibiotic | 7 days
Bacteriological failure, defined as persistent isolation of Staphylococcus aureus with the same phenotype 7 days after or more after treatment onset | 7 days
Need for surgical intervention or other invasive procedures | 30 days
Need for central catheter removal | 30 days
Persistent bacteremia | 30 days
All-cause mortality in ICU and in-hospital | 30 days
Adverse events | 30 days
Durations of fever, assigned antibiotic treatment, mechanical ventilation, ICU and hospital stay | 30 days
Resistance development | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mical Paul, MD, Principal Investigator — Rabin Medical Center; Jihad Bishara, MD, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center; Beilinson Hospital and Davidoff Cancer Center, Petah Tikva

REFERENCES:
- [Derived] Paul M, Bishara J, Yahav D, Goldberg E, Neuberger A, Ghanem-Zoubi N, Dickstein Y, Nseir W, Dan M, Leibovici L. Trimethoprim-sulfamethoxazole versus vancomycin for severe infections caused by meticillin resistant Staphylococcus aureus: randomised controlled trial. BMJ. 2015 May 14;350:h2219. doi: 10.1136/bmj.h2219. PMID 25977146